CLINICAL TRIAL: NCT05743088
Title: COVID-19 Pandemic: Perception, Attitude, and Practices of University Students From Health Sector Faculties.
Brief Title: COVID-19 Pandemic: Perception, Attitude
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nermen Abuelkassem, lecturer, Assiut University
Other Study IDs: covid 19 pandemic
Record Dates: First submitted 2023-02-22; First posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: COVID-19 Pandemic
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: questionnaire — The questionnaire consists of the following parts: socio-demographic data of participants, student perception and attitude towards the COVID-19 pandemic and its consequences, as well as practices of preventive measures in the community.

SUMMARY:
: adherence to preventive control measures is influenced by perception, attitudes and practices toward the disease prevention.

DETAILED DESCRIPTION:
METHODS Study design: A cross-sectional survey study was utilized in which data were collected following the Checklist for Reporting Results of Internet E Surveys (CHERRIES) guidelines during the period from March to July2021.

Study settings and participants The study conducted through an electronic anonymous online survey distributed among students from three health sector faculties (Medicine, Pharmacy, and Nursing) in six Egyptian universities (Cairo, Suez Canal, Tanta, Daria, Aswan, Kufr Elsheikh).

The self-administered online questionnaire was hosted in google form and the link was distributed through official university platforms and informal student groups on social media like Facebook and WhatsApp pages. Representatives of students were also engaged in distributing the questionnaire's link directly to their colleagues from each faculty. A non-randomized convenient sample of 1900 university medical students was included in the study.

Data collection The study questionnaire was developed based on the COVID-19 Rapid Quantitative Assessment Tool as part of the Risk Communication and Community Engagement (RCCE) Action Plan Guidance COVID-19 preparedness and response developed by the China International Famine Relief Commission publication, United Nations Children's Fund (UNICEF) and World Health Organization (WHO) [14]. Most of the questions were in the form of "yes and no" questions except for a few questions with the third "I don't know" option, a five-point rating scale question.

After the tool was developed, the application was tested by the EYI (Egyptian Youth Initiative) executive team at the National Population Council (NPC)/UNICEF to verify, confirm and skip patterns and follow them to guarantee the accuracy of data collection. To ensure the validity and accuracy of the data collected, the investigators settle detailed instructions regarding study objectives for all student counselors who distributed the questionnaire to the subjects in advance. The survey tool automatically verifies that all questions must be filled before submission and cannot be submitted twice.

ELIGIBILITY:
Inclusion creteria university students from health sector faculties

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study conducted through an electronic anonymous online survey distributed among students from three health sector faculties (Medicine, Pharmacy, and Nursing) in six Egyptian universities (Cairo, Suez Canal, Tanta, Daria, Aswan, Kufr Elsheikh).
Sampling Method: Non-Probability Sample
Enrollment: 1990 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
To assess the perceptions, attitude and practices of university students in three health sector faculties (Medicine, Nursing and Pharmacy) from six Egyptian universities towards COVID-19 pandemic prevention. | from march to july 2021

CONTACTS AND LOCATIONS:
Overall Officials: nermen abuelkassem, Lecturer, Principal Investigator — assiut
Locations (1):
- Nermen Mohammed Abuelkassem, Asyut, Egypt